CLINICAL TRIAL: NCT03285646
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Fasinumab in Patients With Moderate-to-Severe Chronic Low Back Pain and Osteoarthritis of the Hip or Knee
Brief Title: Evaluate the Efficacy and Safety of Fasinumab in Patients With Moderate-to-Severe Chronic Low Back Pain and Osteoarthritis of the Hip or Knee
Acronym: FACT CLBP 1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to implementation of an urgent safety measure, enrollment and dosing in R475-PN-1612 was stopped; enrolled participants entered the 20-week safety follow-up
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R475-PN-1612; 2017-001943-12 (EudraCT Number)
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Chronic Low Back Pain; Osteoarthritis
Keywords: Knee; Hip
MeSH Terms: conditions — Osteoarthritis | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasinumab (Experimental): Subcutaneous (SC) every 4 weeks (Q4W)
  Interventions: Drug: Fasinumab
- Placebo (Experimental): SC every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fasinumab — Subcutaneous (SC) every 4 weeks (Q4W)
  Other Names: REGN475
  Arms: Fasinumab
Drug: Placebo — Subcutaneous (SC) every 4 weeks (Q4W)
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of fasinumab in relieving Chronic low back pain (CLBP) as compared to placebo in participants with a clinical diagnosis of moderate-to-severe non-radicular CLBP and Osteoarthritis (OA) of the knee or hip when treated for up to 16 weeks. The secondary objectives of the study are: To evaluate the safety and tolerability of fasinumab compared to placebo when participants with a clinical diagnosis of moderate-to-severe non-radicular CLBP and OA of the knee or hip are treated for up to 16 weeks; To characterize the concentrations of fasinumab in serum over time when participants with a clinical diagnosis of moderate-to-severe non-radicular CLBP and OA of the knee or hip are treated for up to 16 weeks; To evaluate the immunogenicity of fasinumab when treated for up to 16 weeks in participants with a clinical diagnosis of moderate-to-severe non-radicular CLBP and OA of the knee or hip.

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical diagnosis of non-radicular moderate-to-severe CLBP for ≥3 months (prior to screening visit)
2. Clinical diagnosis of OA in at least 1 hip or knee joint based on the American College of Rheumatology Criteria with radiographic evidence of OA (K-L ≥2) at screening
3. History of inadequate relief of CLBP from non-pharmacologic therapy
4. Willing to undergo joint replacement (JR) surgery, if necessary
5. History of regular analgesic medication use
6. History of inadequate pain relief or intolerance to analgesics used for chronic LBP

Key Exclusion Criteria:

1. Patient is not a candidate for MRI
2. History of major trauma or back surgery in the past 6 months prior to the screening visit
3. History or presence of pyriformis syndrome
4. Evidence on baseline lumbar spine magnetic resonance imaging of potentially confounding conditions
5. History or evidence on joint imaging of conditions that may confound joint safety evaluation
6. Evidence or symptoms consistent with autonomic dysfunction (e.g., orthostatic hypotension and/or autonomic symptoms) as defined in the protocol
7. Recent use of longer acting pain medications
8. Other medical conditions that may interfere with participation or accurate assessments during the trial

Note: Other protocol defined Inclusion/ Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (52):
- United States (52):
  - Regeneron Research Site, Phoenix, Arizona
  - Regeneron Research Site, Tucson, Arizona
  - Regeneron Research Site, Anaheim, California
  - Regeneron Research Site, La Mesa, California
  - Regeneron Research Site, North Hollywood, California
  - Regeneron Research Site, San Diego, California
  - Regeneron Research Site, San Marcos, California
  - Regeneron Research Site, Santa Ana, California
  - Regeneron Research Site, Spring Valley, California
  - Regeneron Research Site, Whittier, California
  - Regeneron Research Site, Stamford, Connecticut
  - Regeneron Research Site, Waterbury, Connecticut
  - Regeneron Research Site, Clearwater, Florida
  - Regeneron Research Site, Hialeah, Florida
  - Regeneron Research Site, Jacksonville, Florida
  - Regeneron Research Site, Lauderdale Lakes, Florida
  - Regeneron Research Site, Miami, Florida
  - Regeneron Research Site, Ocoee, Florida
  - Regeneron Research Site, Orlando, Florida
  - Regeneron Research Site, Port Orange, Florida
  - Regeneron Research Site, Sarasota, Florida
  - Regeneron Research Site, Atlanta, Georgia
  - Regeneron Research Site, Columbus, Georgia
  - Regeneron Research Site #1, Marietta, Georgia
  - Regeneron Research Site #2, Marietta, Georgia
  - Regeneron Research Site, Newnan, Georgia
  - Regeneron Research Site, Idaho Falls, Idaho
  - Regeneron Research Site, Chicago, Illinois
  - Regeneron Research Site, Valparaiso, Indiana
  - Regeneron Research Site, West Des Moines, Iowa
  - Regeneron Research Site, Edgewood, Kentucky
  - Regeneron Research Site, New Orleans, Louisiana
  - Regeneron Research Site, Bay City, Michigan
  - Regeneron Research Site, St Louis, Missouri
  - Regeneron Research Site, Lincoln, Nebraska
  - Regeneron Research Site, Las Vegas, Nevada
  - Regeneron Research Site, Berlin, New Jersey
  - Regeneron Research Site, Albuquerque, New Mexico
  - Regeneron Research Site, Hartsdale, New York
  - Regeneron Research Site, New York, New York
  - Regeneron Research Site, High Point, North Carolina
  - Regeneron Research Site, Fargo, North Dakota
  - Regeneron Research Site, Beavercreek, Ohio
  - Regeneron Research Site, Oklahoma City, Oklahoma
  - Regeneron Research Site, Duncansville, Pennsylvania
  - Regeneron Research Site, Rapid City, South Dakota
  - Regeneron Research Site #1, Memphis, Tennessee
  - Regeneron Research Site #2, Memphis, Tennessee
  - Regeneron Research Site, Houston, Texas
  - Regeneron Research Site, Katy, Texas
  - Regeneron Research Site, Plano, Texas
  - Regeneron Research Site, Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for study eligibility across the US. Of the 377 participants screened, 63 met eligibility criteria. The most frequently reported reason for non-randomization was inclusion criteria not met and/or exclusion criteria met (224 participants):139 did not meet inclusion criteria, 86 participants met exclusion criteria.
Pre-assignment Details: The study consisted of a screening period of up to 30 days and a 7 (+3 day) day pre-randomization period during which all pain medication except study-provided rescue medication was discontinued.
Groups:
- Fasinumab-matching Placebo: Participants received fasinumab-matching placebo subcutaneously (SC) every 4 weeks (Q4W) from day 1 through week 12 of the 16 week treatment period. Participants were permitted to use only acetaminophen/paracetamol as rescue medication. The treatment period included both study visits and a phone contact on day 8 (±1 day) up to 16 weeks.
- Fasinumab 3 mg SC Q4W: Participants received fasinumab 3 milligrams (mg) subcutaneously (SC) every 4 weeks (Q4W) from day 1 through week 12 of the 16 week treatment period. Participants were permitted to use only acetaminophen/paracetamol as rescue medication. The treatment period included both study visits and a phone contact on day 8 (±1 day) up to 16 weeks.
Period: Overall Study
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Started | 32 | 31
Completed | 19 | 27
Not Completed | 13 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 10 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Investigator/Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (9.88) | 60.0 (10.52) | 58.8 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 31 | 28 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 15 | 17 | 32
  Black or African American | 15 | 14 | 29
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
Average Daily Low Back Pain Intensity (LBPI) Numerical Rating Scale (NRS) Score [Mean (Standard Deviation); unit: Score on a Scale] — Average daily low back pain (LBP) was assessed on an 11-point numeric rating scale (NRS) and was defined as the average of the non-missing daily LBPI NRS scores for the 7 days before and including nominal visit. Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate higher pain.
  Score on a Scale | 6.66 (1.475) | 6.81 (1.338) | 6.73 (1.400)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in the Average Daily Low Back Pain Intensity (LBPI) Numeric Rating Scale (NRS) Score
Description: Average daily low back pain (LBP) was assessed on an 11-point numeric rating scale (NRS) and was defined as the average of the non-missing daily LBPI NRS scores for the 7 days before and including nominal visit. Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate higher pain.
Time Frame: Week 1, Week 2, Week 4, Week 8, Week 12, Week 16
Population: Number of Participants analyzed = Participants evaluable for this endpoint
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Score on a Scale
  Change from Baseline to Week 1 | -0.73 (1.424) | -1.62 (2.037)
  Change from Baseline to Week 2: number analyzed (Participants) | 29 | 31
  Change from Baseline to Week 2 | -0.98 (1.588) | -2.15 (2.067)
  Change from Baseline to Week 4: number analyzed (Participants) | 28 | 29
  Change from Baseline to Week 4 | -1.28 (1.878) | -2.64 (2.038)
  Change from Baseline to Week 8: number analyzed (Participants) | 20 | 21
  Change from Baseline to Week 8 | -1.21 (1.568) | -2.82 (1.963)
  Change from Baseline to Week 12: number analyzed (Participants) | 9 | 13
  Change from Baseline to Week 12 | -2.12 (1.582) | -3.18 (2.046)
  Change from Baseline to Week 16: number analyzed (Participants) | 2 | 7
  Change from Baseline to Week 16 | -0.77 (1.943) | -2.32 (1.367)

2. Secondary Outcome: Change From Baseline to Week 16 in the Roland Morris Disability Questionnaire (RMDQ) Total Score
Description: The RMDQ is a self-administered, health status measure for lower back pain (LBP). It measures pain and function using 24 items describing limitations to everyday life that can be caused by LBP. The score of the RMDQ is the total number of items checked from a minimum of 0 (no disability) to a maximum of 24 (maximum disability), where lower scores are indicative of better function.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16
Population: Number of Participants Analyzed = Participants evaluable for this endpoint
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Score on a Scale
  Change from Baseline to Week 2: number analyzed (Participants) | 27 | 24
  Change from Baseline to Week 2 | -2.70 (5.120) | -2.54 (4.836)
  Change from Baseline to Week 4: number analyzed (Participants) | 24 | 23
  Change from Baseline to Week 4 | -1.92 (4.529) | -3.09 (3.884)
  Change from Baseline to Week 8: number analyzed (Participants) | 19 | 17
  Change from Baseline to Week 8 | 0.37 (4.487) | -4.18 (5.015)
  Change from Baseline to Week 12: number analyzed (Participants) | 6 | 9
  Change from Baseline to Week 12 | 0.83 (3.061) | -3.33 (4.301)
  Change from Baseline to Week 16: number analyzed (Participants) | 1 | 4
  Change from Baseline to Week 16 | -1.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants | -5.75 (3.948)

3. Secondary Outcome: Change From Baseline to Week 16 in Patient Global Assessment (PGA) of Low Back Pain (LBP) Score
Description: The PGA of LBP is a participant assessed 5 point Likert scale of LBP ranging from 1-5 where 1 = very well; 2 = well; 3 = fair; 4 = poor; and 5 = very poor.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16
Population: Number of Participants Analyzed = Participants evaluable for this endpoint
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Score on a Scale
  Change from Baseline to Week 2: number analyzed (Participants) | 27 | 29
  Change from Baseline to Week 2 | -0.44 (0.751) | -0.76 (0.786)
  Change from Baseline to Week 4: number analyzed (Participants) | 25 | 25
  Change from Baseline to Week 4 | -0.60 (0.957) | -1.04 (0.676)
  Change from Baseline to Week 8: number analyzed (Participants) | 20 | 20
  Change from Baseline to Week 8 | -0.55 (0.945) | -1.10 (1.021)
  Change from Baseline to Week 12: number analyzed (Participants) | 7 | 10
  Change from Baseline to Week 12 | -0.57 (1.134) | -1.00 (1.333)
  Change from Baseline to Week 16: number analyzed (Participants) | 1 | 4
  Change from Baseline to Week 16 | 0.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants | -0.75 (0.500)

4. Secondary Outcome: Number of Participants Achieving ≥30% Reduction From Baseline to Week 16 in Average Daily LBPI NRS Score
Description: as for outcome 1
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Participants | 12 | 21

5. Secondary Outcome: Change From Baseline to Week 16 in the Brief Pain Inventory-Short Form (BPI-sf) Pain Interference Score
Description: The BPI-sf is a self-administered questionnaire for participants to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function. With a recall period of 24 hours, the questionnaire contains the front and back body diagrams, the 4 pain severity items and 7 pain interference items rated on 0-10 scale; total interference score ranges from 0-10 (0, does not interfere; 10 completely interferes), and the question about percentage of pain relief by analgesics. The BPI pain interference is typically scored as the mean of the 7 interference items.
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16
Population: Number of Participants Analyzed = Participants evaluable for this endpoint
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Score on a Scale
  Change from Baseline to Week 2: number analyzed (Participants) | 27 | 29
  Change from Baseline to Week 2 | -1.55 (2.306) | -1.94 (2.255)
  Change from Baseline to Week 4: number analyzed (Participants) | 25 | 25
  Change from Baseline to Week 4 | -1.49 (2.390) | -2.15 (2.157)
  Change from Baseline to Week 8: number analyzed (Participants) | 20 | 20
  Change from Baseline to Week 8 | -1.31 (2.119) | -2.70 (2.774)
  Change from Baseline to Week 12: number analyzed (Participants) | 7 | 10
  Change from Baseline to Week 12 | -1.63 (2.096) | -1.84 (1.978)
  Change from Baseline to Week 16: number analyzed (Participants) | 1 | 4
  Change from Baseline to Week 16 | -1.14 (NA) — Standard deviation could not be calculated due to insufficient number of participants | -1.29 (3.017)

6. Secondary Outcome: Number of Adjudicated Arthropathy (AA) Events
Description: Adjudicated arthropathy (AA) is a composite term that encompasses the following conditions: Rapidly progressive OA type 1 and 2, Subchondral insufficiency fractures, and Primary Osteonecrosis. AAs were also evaluated to determine if they met Destructive Arthropathy criteria.
Time Frame: Up to Week 36
Measure: Number; unit: Adjudicated Arthropathy (AA) Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Adjudicated Arthropathy (AA) Events | 0 | 2

7. Secondary Outcome: Number of Adjudicated Arthropathy (AA) Events Meeting Destructive Arthropathy (DA) Criteria
Description: Destructive arthropathy (DA) is a unique clinical form of rapidly destructive arthropathy over and above that seen in the normal progression of OA. DA criteria can be associated with Rapidly Progressive Osteoarthritis type 2, Subchondral Insufficiency fracture, and Primary Osteonecrosis.
Time Frame: Up to Week 36
Measure: Number; unit: Destructive Arthropathy (DA) Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Destructive Arthropathy (DA) Events | 0 | 0

8. Secondary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAEs) are defined as those that are not present at baseline or represent the exacerbation of a pre-existing condition during the on-treatment period.
Time Frame: Up to Week 16
Measure: Number; unit: Treatment-Emergent Adverse Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Treatment-Emergent Adverse Events | 33 | 14

9. Secondary Outcome: Number of Sympathetic Nervous System (SNS) Dysfunction Events
Description: Potential events of sympathetic nervous system (SNS) dysfunction were monitored throughout the study through physical examination, AE reporting, assessment of orthostatic hypotension, and the Survey of Autonomic Symptoms. Sympathetic nervous system dysfunction was diagnosed after consultation with an appropriate specialist, such as a neurologist and/or cardiologist.
Time Frame: Up to Week 36
Measure: Number; unit: Sympathetic NS Dysfunction Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Sympathetic NS Dysfunction Events | 0 | 0

10. Secondary Outcome: Number of Peripheral Sensory Adverse Events (AEs) That Require a Neurology Consultation
Description: Any peripheral sensory AE (eg, paraesthesia and hypoaesthesia) that required a neurology consultation.
Time Frame: Up to Week 36
Measure: Number; unit: Peripheral Sensory Adverse Events (AEs)
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Peripheral Sensory Adverse Events (AEs)
  Hypoaesthesia events | 1 | 0
  Paraesthesia events | 1 | 0

11. Secondary Outcome: Number of All-Cause Joint Replacement (JR) Surgery Events
Description: All joint replacement surgery events regardless of cause.
Time Frame: Up to Week 36
Measure: Number; unit: Joint Replacement (JR) Surgery Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Joint Replacement (JR) Surgery Events | 2 | 1

12. Secondary Outcome: Number of Joint Replacement (JR) Surgery Events Reported at Telephone Survey After Last Dose of Study Drug
Description: An end of study phone contact was conducted approximately 52 weeks following the last dose of study drug (week 12) to evaluate the number of participants who had undergone or were scheduled for JR surgery.
Time Frame: Up to Week 64
Measure: Number; unit: Joint Replacement (JR) Surgery Events
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 32 | 31
Joint Replacement (JR) Surgery Events | 0 | 0

13. Secondary Outcome: Number of Participants With at Least One Positive Anti-Drug Antibody (ADA) Assay
Description: Samples for Anti-Drug Antibody (ADA) evaluation were collected at baseline and at subsequent study visits. ADA variables include ADA status (+ or -) and titer as follows: Total participants negative in the ADA assay at all time points analyzed. Pre-existing immunoreactivity - positive response at baseline with all post-dose results negative, or a positive response at baseline with all post-dose responses less than 9-fold over baseline titer levels. Treatment emergent - post-dose positive result when baseline results were negative. Persistent - A positive result detected in at least 2 consecutive post baseline samples separated by at least a 16-week post baseline period, with no negative results in-between. Indeterminate - A positive result at the last collection time point analyzed only. Transient - Not persistent or indeterminate regardless of any missing samples. Treatment boosted - any post-dose positive result at least 9-fold over the baseline level when baseline is positive.
Time Frame: 16 Weeks
Population: Anti-Drug Antibody (ADA) analysis set: All treated participants who received any study drug or placebo (safety analysis set) and had at least one non-missing anti-drug antibody result following the first dose of study drug or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 31 | 31
Participants
  Negative/Pre-Existing | 31 | 31
  Treatment Boosted | 0 | 0
  Treatment-Emergent | 0 | 0
  Treatment-Emergent: Persistent | 0 | 0
  Treatment-Emergent: Transient | 0 | 0
  Treatment-Emergent: Indeterminate | 0 | 0

14. Secondary Outcome: Serum Concentration of Functional Fasinumab Over Time
Description: Summary of mean concentration of functional fasinumab are presented by nominal time point.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 16
Population: Number of Participants Analyzed = Participants evaluable for this endpoint
Measure: Mean (Standard Deviation); unit: Milligram per Liter (mg/L)
Arm/Group | Fasinumab 3 mg SC Q4W
Number analyzed (Participants) | 31
Milligram per Liter (mg/L)
  Baseline | 0 (0)
  Week 2: number analyzed (Participants) | 23
  Week 2 | 0.262 (0.0992)
  Week 4: number analyzed (Participants) | 25
  Week 4 | 0.176 (0.0679)
  Week 8: number analyzed (Participants) | 18
  Week 8 | 0.247 (0.130)
  Week 16: number analyzed (Participants) | 3
  Week 16 | 0.192 (0.0932)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 24 weeks post the last dose of study drug (up to week 36)
Description: Reported adverse events (AEs) are AEs that developed/worsened from the time of the first administration of study drug until the end of the follow up period (week 36)
Arm/Group | Fasinumab-matching Placebo | Fasinumab 3 mg SC Q4W
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/32 | 2/31
Other Adverse Events (participants affected / at risk) | 14/32 | 4/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasinumab-matching Placebo (N=32) | Fasinumab 3 mg SC Q4W (N=31)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasinumab-matching Placebo (N=32) | Fasinumab 3 mg SC Q4W (N=31)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (4)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment and study drug administration was stopped due to an urgent safety measure. As a result the small number of participants enrolled in this study limited the interpretability of the efficacy results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT03285646/Prot_002.pdf
  • Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT03285646/SAP_003.pdf